CLINICAL TRIAL: NCT03212924
Title: Evaluation of Listening Effort With Pupillometry in Cochlear Implant Users
Brief Title: Listening Effort in Cochlear Implant Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIC_13
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Sensorineural Hearing Loss; Cochlear Hearing Loss
Keywords: cochlear implant; Listening effort; pupillometry
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Noise; Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pupillometry (Experimental): Measure of pupil dilatation while listening to speech (monosyllabic words) in quiet and in noise.
  Evaluation of speech comprehension in quiet
  Evaluation of speech comprehension in noise
  Measure of cognitive functions with the MOCA (Montreal Cognitive Assessment)
  Auto evaluation of listening effort in quiet
  Auto evaluation of listening effort in noise
  Interventions: Behavioral: Pupillometry; Behavioral: Evaluation of speech comprehension in quiet; Behavioral: Evaluation of speech comprehension in noise; Behavioral: MOCA; Behavioral: auto evaluation of listening effort in quiet; Behavioral: auto evaluation of listening effort in noise

INTERVENTIONS:
Behavioral: Pupillometry — Measure of pupil dilatation simultaneously to the evaluation of speech intelligibility. The variation of the pupil size is monitored during the presentation of speech stimuli in quiet and in the presence of a background noise.
Behavioral: Evaluation of speech comprehension in quiet — Three lists of 17 monosyllabic words (Lafon) are presented in quiet at 65 dB SPL. Listeners have to repeat what they understood. The results correspond to the percent of phonemes correctly identified.
Behavioral: Evaluation of speech comprehension in noise — Three lists of 17 monosyllabic words (Lafon) are presented in a wide band noise at 65 dB SPL with a SNR (signal to noise ratio) of +10 dB. Listeners have to repeat what they understood. The results correspond to the percent of phonemes correctly identified.
Behavioral: MOCA — The Montreal Cognitive Assessment (MoCA) is a screening instrument to detect cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The time to administer the MoCA is approximately 10 minutes. The total possible score is 30 points. The test suggests the existence of a cognitive impairment if the participant scores less than 26 points. The test is presented on a single sheet of paper.
  Other Names: Montreal Cognitive Assessment
Behavioral: auto evaluation of listening effort in quiet — The participant has to represent, on a continuous line, the amount of listening effort he used when listening to the monosyllabic words presented in quiet. A score from 0 (no listening effort) to 10 (effort maximum) is extracted from his response.
  Other Names: VAS (visual analog scale) in quiet
Behavioral: auto evaluation of listening effort in noise — The participant has to represent, on a continuous line, the amount of listening effort he used when listening to the monosyllabic words presented in the background noise. A score from 0 (no listening effort) to 10 (effort maximum) is extracted from his response.
  Other Names: VAS (visual analog scale) in noise

SUMMARY:
Listening with a cochlear implant remains difficult and most listeners will report high levels of listening effort.The present study is a "pilot" aiming to evaluate listening effort for cochlear implant users. The listening effort is measured with pupillometry, by monitoring the variations of pupil size in response to different stimuli. The size of the pupil is known to increase with the listening effort. The listening effort is evaluated in two different situation: speech perception in quiet and speech perception in noise. The pupillometry measures will be compared for the two listening conditions. Moreover, the study will evaluate the relationship between objective (pupil dilatation) and subjective measures (auto evaluation) of listening effort, and between speech comprehension, cognitive abilities and listening effort.

DETAILED DESCRIPTION:
Nowadays, cochlear implants (CI) are successfully used to rehabilitate severe to profound sensorineural hearing loss. Most CI users can understand speech in quiet, but comprehension scores drop in the presence of background noise and in adverse conditions. Listening with a cochlear implant remains very demanding and most listeners report high levels of listening effort. The aim of current auditory prostheses and cochlear implants is not only restore speech understanding, but also to restore all the cognitive functions that are associated to a listening task (e.g., memory, executive functions, attention). Evaluating the listening effort is a new way to assess the efficiency of the hearing aids or cochlear implants. The listening effort indicates the amount of cognitive resources that are dedicated to a listening task; it evaluates also the cognitive resources remaining available for the other cognitive functions. The present study is a "pilot" aiming to evaluate listening effort for cochlear implant users. The listening effort is measured with pupillometry, i. e. by measuring the pupil dilatation in response to different stimuli. The size of the pupil is known to increase with the listening effort. The listening effort is evaluated in two different situation: speech perception in quiet and speech perception in noise. Speech comprehension is measured for the two listening conditions and cognitive functions are assessed by the MOCA (Montreal Cognitive Assessment). In addition, the subjects are asked to subjectively evaluate the amount of listening effort they used in each listening situation. The pupillometry measures will be compared for the two listening conditions. Moreover, the study will evaluate the relationship between objective (pupil dilatation) and subjective measures (self evaluation) of listening effort, and between speech comprehension, cognitive abilities and listening effort.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* Native French speaker or fluent French speaker
* Patient already fitted with one or two cochlear implants Oticon Medical
* Can correctly identify at least 10 % of the words in monosyllabic Lafon lists in quiet
* Normal or corrected to normal vision

Exclusion Criteria:

* vulnerable patients (kids, pregnant women, persons under guardianship)
* No Social security affiliation
* blindness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2018-03-27 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
Pupil dilatation (mm) | 1 hour
  The listening effort while listening to speech stimuli is estimated by measuring the pupil size relative to a baseline. Measures of pupil dilatation are compared between quiet and noisy conditions (+ 10 SNR: signal to noise ratio).
Amplitude of peak of pupil dilatation | 1 hour
  The listening effort while listening to speech stimuli is estimated by measuring the pupil size relative to a baseline. The peak is defined as the point in time where the maximum of pupil dilatation occurs. The amplitude of the peak of dilatation is compared between quiet and noisy conditions (+ 10 SNR: signal to noise ratio).
Latency of peak of pupil dilatation (ms) | 1 hour
  The listening effort while listening to speech stimuli is estimated by measuring the pupil size relative to a baseline. The peak is defined as the point in time where the maximum of pupil dilatation occurs. The latency of the peak of dilatation is compared between quiet and noisy conditions (+ 10 SNR: signal to noise ratio).

SECONDARY OUTCOMES:
Speech intelligibility in quiet | 30 mins simultaneously to pupillometry measures
  percentage of phonemes correctly identify when the speech stimuli (monosyllabic words of Lafon) are presented in quiet at 65 dB SPL
Speech intelligibility in noise | 30 mins simultaneously to pupillometry measures
  percentage of phonemes correctly identify when the speech stimuli (monosyllabic words of Lafon) are presented in a wide band noise at 65 dB SPL with a +10 dB SNR (signal to noise ratio)
MOCA (Montreal Cognitive assessment) | 15 mins
  Score at the MOCA. The maximum score is 30. The test suggests the existence of a cognitive impairment if the score is lower than 26.
VAS quiet | 1 min
  Auto evaluation of the listening effort in quiet with Visual Analog Scale. The participant has to indicate, on a continuous line, the listening effort used in the quiet condition. A score from 0 (no effort) to 10 (maximum effort) is extracted from the VAS.
VAS noise | 1 min
  Auto evaluation of the listening effort in quiet with Visual Analog Scale. The participant has to indicate, on a continuous line, the listening effort used in the noise condition. A score from 0 (no effort) to 10 (maximum effort) is extracted from the VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Mosnier, MD, Principal Investigator — Hôpital Pitié Sapêtrière - APHP
Locations (1):
- Hôpital Pitié Salpêtrière - APHP, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kramer SE, Teunissen CE, Zekveld AA. Cortisol, Chromogranin A, and Pupillary Responses Evoked by Speech Recognition Tasks in Normally Hearing and Hard-of-Hearing Listeners: A Pilot Study. Ear Hear. 2016 Jul-Aug;37 Suppl 1:126S-35S. doi: 10.1097/AUD.0000000000000311. PMID 27355762
- [Result] Steel MM, Papsin BC, Gordon KA. Binaural fusion and listening effort in children who use bilateral cochlear implants: a psychoacoustic and pupillometric study. PLoS One. 2015 Feb 10;10(2):e0117611. doi: 10.1371/journal.pone.0117611. eCollection 2015. PMID 25668423
- [Result] Winn MB, Edwards JR, Litovsky RY. The Impact of Auditory Spectral Resolution on Listening Effort Revealed by Pupil Dilation. Ear Hear. 2015 Jul-Aug;36(4):e153-65. doi: 10.1097/AUD.0000000000000145. PMID 25654299
- [Result] Koelewijn T, Zekveld AA, Festen JM, Kramer SE. Pupil dilation uncovers extra listening effort in the presence of a single-talker masker. Ear Hear. 2012 Mar-Apr;33(2):291-300. doi: 10.1097/AUD.0b013e3182310019. PMID 21921797
- [Result] Zekveld AA, Kramer SE. Cognitive processing load across a wide range of listening conditions: insights from pupillometry. Psychophysiology. 2014 Mar;51(3):277-84. doi: 10.1111/psyp.12151. Epub 2014 Feb 9. PMID 24506437
- [Result] Zekveld AA, Heslenfeld DJ, Johnsrude IS, Versfeld NJ, Kramer SE. The eye as a window to the listening brain: neural correlates of pupil size as a measure of cognitive listening load. Neuroimage. 2014 Nov 1;101:76-86. doi: 10.1016/j.neuroimage.2014.06.069. Epub 2014 Jul 3. PMID 24999040
- [Result] Zekveld AA, Kramer SE, Festen JM. Cognitive load during speech perception in noise: the influence of age, hearing loss, and cognition on the pupil response. Ear Hear. 2011 Jul-Aug;32(4):498-510. doi: 10.1097/AUD.0b013e31820512bb. PMID 21233711
- [Result] Zekveld AA, Kramer SE, Festen JM. Pupil response as an indication of effortful listening: the influence of sentence intelligibility. Ear Hear. 2010 Aug;31(4):480-90. doi: 10.1097/AUD.0b013e3181d4f251. PMID 20588118
- [Result] Pals C, Sarampalis A, Baskent D. Listening effort with cochlear implant simulations. J Speech Lang Hear Res. 2013 Aug;56(4):1075-84. doi: 10.1044/1092-4388(2012/12-0074). Epub 2012 Dec 28. PMID 23275424